CLINICAL TRIAL: NCT01614561
Title: CEPHEUS Centralized Pan-Levant Survey on the Undertreatment of Hypercholesterolemia NIS-LT-CRE-2010/01 Version 1.0
Brief Title: An Observational Study Evaluating Cholesterol Levels in Patients on Cholesterol Lowering Drugs in Jordan and Lebanon
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-LT-CRE-2010/01
Record Dates: First submitted 2012-06-01; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: High Blood Cholesterol
Keywords: Hypercholesterolemia; Lipid lowering drugs; Cholesterol level in blood; Target cholesterol levels guidelines for the management of high blood cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood specimens, serum, non-retained
Oversight: Data Monitoring Committee: No

SUMMARY:
This was a multicenter survey of patients who were on lipid -lowering pharmacological treatment in 2 Levant countries namely Jordan and Lebanon. The purpose is to study the effects of cholesterol lowering drugs on the blood cholesterol levels of patients in Jordan and Lebanon.

Data collected from each patient took place at a single visit. Each participating doctor filled the investigator questionnaire on his/her experience and perception of the management of the hypercholesterolemia of his/her patients. Each doctor was asked to indicate his/her general attitude on the diagnosis of hypercholesterolemia, the existing guidelines and goals and the various treatment options for high cholesterol in blood.

Before being assessed by the investigator, patients recorded, on the patient questionnaire, their awareness of high blood cholesterol , their current lipid-lowering treatment schedule, their understanding of their condition and compliance in taking the medications on time.

The investigators completed a Patient Record Form (PRF) with the patient's basic information, cardiovascular risk factors and the cardiovascular medical history, current lipid lowering drug treatment and the reason for the current therapy.

A blood sample under fasting condition was drawn from each subject. A central laboratory in Jordan received all samples. Every sample was analyzed for its cholesterol blood level, fasting sugar level and hemoglobin A1C levels.

DETAILED DESCRIPTION:
CEPHEUS Centralized Pan-Levant Survey on the Undertreatment of Hypercholesterolemia NIS-LT-CRE-2010/01 Version 1.0

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with high cholesterol blood levels willing to participate in the study
* Patients must be on cholesterol lowering medications for three months with no dose change for six weeks

Exclusion Criteria:

* Patients not on cholesterol lowering medications or on medications for less than three months
* Any medication dose change in six weeks prior to their visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending out patient clinics in Jordan and Lebanon
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects achieving the LDL-C goals, according to the NCEP ATP III / updated 2004 NCEP ATP III guidelines, in Jordan and Lebanon | 5 months- One visit only, no follow up visits

SECONDARY OUTCOMES:
Number and percentage of subjects achieving LDL-C goals according to the NCEP ATP III / 2004 updated NCEP ATP III guidelines, for several subject subsets | 5 months- One visit only, no follow up visits
Number and percentage of subjects achieving the LDL-C goals, according to the Third Joint European Task Force guidelines, overall and for several subject subsets | 5 months- One visit only, no follow up visits
Number and percentage of subjects achieving the non HDL-C goals according to the NCEP ATP III / updated 2004 NCEP ATP III / national guidelines (<130 mg/dL), in the following sub-population: patients with fasting triglycerides >200 mg/dL. | 5 months- One visit only, no follow up visits
Achievement of LDL-C goals, according to the Third Joint European Task Force TJETF / NCEP ATP III / 2004 updated NCEP ATP III guidelines, and patient and physician variables. Assessed using Multivariate logistic regression mode | 5 months- One visit only, no follow up visits
Physician characteristics associated with the allocation of treatment regimen. | 5 months- One visit only, no follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hammoudeh, MD, Principal Investigator — Istishari Hospital Amman